CLINICAL TRIAL: NCT03844711
Title: Transcutaneous Electrical Diaphragmatic Stimulation and Inspiratory Muscle Training in Healthy Individuals and Patients With Chronic Obstructive Pulmonary Disease Exacerbated
Brief Title: Transcutaneous Electrical Diaphragmatic Stimulation and Inspiratory Muscle Training in Patients With COPD Exacerbated
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-0078
Record Dates: First submitted 2019-01-26; First posted 2019-02-18 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Electrical Stimulation; Respiratory Muscle Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous electrical diaphragmatic stimulation (TEDS) (Experimental): For transcutaneous electrical diaphragmatic stimulation, surface electrodes will be used that will be positioned at the transcutaneous motor points of the diaphragm.
  Interventions: Other: Transcutaneous electrical diaphragmatic stimulation (TEDS); Other: Conventional physiotherapy
- Inspiratory Muscle training (IMT) (Experimental): The training will start with a minimum load of 50% and will be progressed until reaching 60% of the PImax.
  Interventions: Other: Inspiratory Muscle Training (IMT); Other: Conventional physiotherapy
- Conventional physiotherapy (Active Comparator): The protocol of physiotherapy by the physiotherapists of HCPA will be twice a day and consists of ventilatory exercises, bronchial hygiene techniques, passive, active-assisted or active exercises for upper and lower limbs, and resistance exercises.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Transcutaneous electrical diaphragmatic stimulation (TEDS) — * Stage I: In the first day (group 1) the parameters will be with 30 Hz frequency and the second day (group 2) will be with 80 Hz, with one-day interval between interventions. The TEDS will be applied with symmetrical biphasic pulsed current, pulse width 0.4 ms, rise time of 1 second (s), 1s lift, 2 s descent, maintaining respiratory rate of 15 rpm, intensity required to obtain visible muscle contraction, for 20 minutes or until muscle fatigue.
  * Stage II and III:The TEDS will be applied with symmetrical biphasic pulsed current, the parameters will be with 30 Hz frequency, pulse width 0.4 ms, rise time of 1 second (s), 1s lift, 2 s descent, maintaining respiratory rate of 15 rpm, intensity required to obtain visible muscle contraction, for 20 minutes or until muscle fatigue.
  Other Names: Transcutaneous electrical diaphragmatic stimulation
  Arms: Transcutaneous electrical diaphragmatic stimulation (TEDS)
Other: Inspiratory Muscle Training (IMT) — - Stage II and III: The training will start with a minimum load of 50% and will be progressed until reaching 60% of the PImax. Inspiratory muscle training will start with a minimum load of 50% and progress to 60% of the MIP. The patients will perform daily training, being two sets of 30 breaths, one in the morning and one in the afternoon.
  Arms: Inspiratory Muscle training (IMT)
Other: Conventional physiotherapy — - Stage III: It consists of ventilatory exercises, bronchial hygiene techniques, passive, active-assisted or active exercises for upper and lower limbs, and resistance exercises.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by chronic airflow limitation, a qualification of impairment of respiratory muscle function, including hyperinflation and muscle weakness. Thus, pulmonary rehabilitation is indicated for patients and is recommended for even the most severe cases. However some patients do not conclude conventional rehabilitation protocols, due to exercise intolerance, are then an electrical estimation and muscle training respiratory adjuvant treatments for patients. and little has been explored about the effects and methodologies of using transcutaneous electrical diaphragmatic stimulation (TEDS) in healthy subjects. The objective of this study on stage I is to evaluate the acute effect of transcutaneous electrical diaphragmatic stimulation on respiratory muscle strength, cardiac variability, thickness, resistance, mobility and diaphragmatic activation comparing different frequencies of electrical stimulation in healthy individuals. The objective of this study on stage II is to evaluate the effects of transcutaneous electrical diaphragmatic stimulation, compared to inspiratory muscle training on respiratory muscle strength, security of the technics, thickness and diaphragmatic function in healthy individuals.The objective of this study on stage III is to evaluate the effects of transcutaneous electrical diaphragmatic stimulation, compared to IMT on respiratory muscle strength, lung function, thickness and diaphragmatic function in patients with exacerbated chronic obstructive pulmonary disease. The study was approved by the Research Ethics Committee of the Hospital de Clinicas of Porto Alegre (CAEE: 80271517.2.0000.5327).

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by chronic airflow limitation, a qualification of impairment of respiratory muscle function, including hyperinflation and muscle weakness. Thus, pulmonary rehabilitation is indicated for patients and is recommended for even the most severe cases. However some patients do not conclude conventional rehabilitation protocols, due to exercise intolerance, are then an electrical estimation and muscle training respiratory adjuvant treatments for patients. and little has been explored about the effects and methodologies of using TEDS in healthy subjects. The objective of this study on stage I is to evaluate the acute effect of transcutaneous electrical diaphragmatic stimulation on respiratory muscle strength, cardiac variability, thickness, resistance, mobility and diaphragmatic activation comparing different frequencies of electrical stimulation in healthy individuals.The objective of this study on stage II is to evaluate the effects of transcutaneous electrical diaphragmatic stimulation, compared to inspiratory muscle training on respiratory muscle strength, security of the technics, thickness and diaphragmatic function in healthy individuals.The objective of this study on stage III is to evaluate the effects of transcutaneous electrical diaphragmatic stimulation, compared to inspiratory muscle training on respiratory muscle strength, lung function, thickness and diaphragmatic function in patients with exacerbated chronic obstructive pulmonary disease. Methods: The Stage I is a cross-over Randomized Controlled Trial (RCT) in the first stage of this research, which will be performed at the Exercise Research Laboratory (LAPEX) of the School of Physical Education, Physiotherapy and Dance of the Universidade Federal do Rio Grande do Sul, the Stage II and is a randomized crossover clinical trial, to be performed at the Exercise Physiology Laboratory (LAFIEX) of Hospital de Clínicas de Porto Alegre (HCPA). Healthy individuals aged between 20 and 60 years, fully aware and cooperative, randomized into two groups will be included: one group that will perform TEDS and another that will perform IMT in a single session. TEDS will be applied with symmetrical biphasic pulsed current, frequency 30 Hertz (Hz), pulse width 0.5 ms, rise time of 1 second, sustain of 1s, descent of 2 s, maintaining respiratory rate of 15 rpm, intensity necessary to obtain muscle contraction visible, for 30 minutes or until muscle fatigue, daily. The IMT will be performed with the PowerBreath device with a charge of 50-60% of the PImax, for 30 breaths and Stage III will be an RCT, which will be performed at the Hospitalization Units of Hospital de Clinicas de Porto Alegre (HCPA). In the first stage only healthy individuals will be included, who will be randomized to TEDS, in the first day (group 1) the parameters will be with 30 hertz (Hz) frequency and the second day (group 2) will be with 80 Hz, with one-day interval between interventions. The TEDS will be applied with symmetrical biphasic pulsed current, pulse width 0.4 ms, rise time of 1 second (s), 1s lift, 2 s descent, maintaining respiratory rate of 15 breaths per minute, intensity required to obtain visible muscle contraction, for 20 minutes or until muscle fatigue. In this stage, heart rate variability, thickness and diaphragmatic mobility by ultrasonography, diaphragmatic activation by electromyography, inspiratory muscle endurance with powerbreath, and respiratory muscle strength by manovacuometry, before and at the end of treatment, the following variables will be measured. In the second stage patients with COPD (GOLD III and IV) hospitalized for exacerbation of the disease, who will be randomized into three groups: one group that will perform TEDS, another will perform IMT and a third group that will only perform conventional physiotherapy. The TEDS will be applied with symmetrical biphasic pulsed current, frequency 30 Hz, pulse width 0.4 ms, rise time of 1 second, sustain of 1s, decrease of 2 s, maintaining respiratory rate (RR) of 15 breaths per minute (rpm), intensity required to obtain visible muscle contraction for 20 minutes or even muscle fatigue daily. The IMT will be performed with the Power Breath device with load referring to 30-60% of PImax, during 30 breaths daily. Conventional physical therapy will be HCPA standard. In this stage, before and at the end of treatment, the following variables will be measured: respiratory muscle strength through manovacuometry, pulmonary function through spirometry, diaphragmatic thickness through echocardiography, diaphragmatic function through respiratory electroneuromyography, Body Mass-Index, Airflow Obstruction, Dyspnea and Exercise Capacity (BODE) Index with mass index (BMI), functional capacity through the six-minute walk test, dyspnoea by the Borg Scale and Medical Research Council (MRC) Scale, cardiovascular variables and time of hospitalization through the electronic medical record. The interventions will be carried out from the patient's hospitalization to the hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Stage I: Healthy adults between 18 and 60 years old; Intense phrenic nerve.
* Stage II: Healthy adults between 20 and 60 years old; Intense phrenic nerve.
* Stage III: Adults between 40 and 80 years old; Smoking more than 10 pack-years; Clinical diagnosis of COPD, GOLD 3 and 4; Patients admitted for severe COPD exacerbation (appearance or worsening of dyspnea, appearance or worsening of cough and appearance or increase in sputum that may be purulent), two of which must be present to characterize exacerbation; Intense phrenic nerve.

Exclusion Criteria (all stages):

* Unstable ventricular arrhythmia;
* Unstable angina; Aortic stenosis;
* Uncontrolled systemic arterial hypertension;
* Epilepsy;
* Undergoing hemodialysis;
* Fever and / or infectious disease;
* Neoplasms;
* Pacemaker;
* At the time of the intervention:
* Oxygen saturation below 90%;
* Obese patients;
* Refuse to participate in the survey.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-16 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength - maximum expiratory pressure (MEP) | One week
  Performed through a manometer in step cmH2O, of the brand Globalmed model MV300. Maximum expiratory pressure.
Respiratory muscle strength - maximum inspiratory pressure (MIP) | One week
  Performed through a manometer in step cmH2O, of the brand Globalmed model MV300. Maximum inspiratory pressure.
Pulmonary function - forced expiratory volume in the first second | One week
  Pulmonary function through spirometry, that allows to measure forced expiratory volume in the first second. It's the maximum expired volume at the first second of an maximum expiration.
Pulmonary function - forced vital capacity | One week
  Pulmonary function through spirometry. Spirometry allows to measure forced vital capacity. It's the air volume expired, quickly, after an inspiration deep maximum.
Diaphragm muscle thickness | One week
  Performed through a Portable Ultrasound System (VIVID i®, GE) with a linear arrangement probe (60 mm, 7.5 Megahertz (MHz) - VIVID i®, GE).
Diaphragm muscle mobility | One week
  Performed through a Portable Ultrasound System (VIVID i®, GE) with a linear arrangement probe (60 mm, 7.5 MHz - VIVID i®, GE).
Electromyography of the diaphragm muscle - Diaphragm Muscle Activation | One week
  Performed through a Portable Electromyograph System (EMG System Brasil Ltda, São José dos Campos) with surface electrodes.
Lower Limb Strength - Test Sit to Stand (STS) | One week
  In the measurements, the subjects mill be asked to stand up from a sitting position and then to sit down 5 times as fast as possible. The STS time will be recorded using a stopwatch to the nearest 10th of a second. The timerequired will be accounted for to perform a 5-time-repeated test on a chair.

SECONDARY OUTCOMES:
Body composition measure (BMI) | One week
  Evaluate the weight of a person in relation to their height.
Dyspnea - Modified Medical Research Council (MRC scale) | One week
  Measure of the subjective sensation of dyspnea.
Dyspnea - BORG scale | One week
  Measure of the subjective sensation of dyspnea. This is a scale that asks you to rate the difficulty of your breathing. It starts at number0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal
Exercise capacity - 6-min walk test (6MWT) | One week
  Distance traveled on the 6MWT.
Systolic blood pressure (SBP) | One week
  Measures the pressure in your blood vessels when your heart beats. Will be measured during each session, using the monitors available on the floors of the HCPA.
Diastolic blood pressure (DBP) | One week
  Measures the pressure in your blood vessels when your heart rests between beats. Will be measured during each session, using the monitors available on the floors of the HCPA.
Heart rate (HR) | One week
  Is the speed of the heartbeat measured by the number of contractions (beats) of the heart per minute (bpm). Will be measured during each session, using the monitors available on the floors of the HCPA.
Respiratory Rate (RR) | One week
  Is the number of breaths you take per minute. Will be measured during each session, using the monitors available on the floors of the HCPA.
Oxygen Saturation (SpO2) | One week
  Is a measurement of how much oxygen the red blood cells in the body's arteries are carrying. Will be measured during each session, using the monitors available on the floors of the HCPA.
Length of hospital stay | One week
  Of the patient's electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Graciele Sbruzzi, Doctor, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No